CLINICAL TRIAL: NCT06843980
Title: Evaluation of the MISHA® Knee System for Symptom Relief in Subjects With Medial Knee Osteoarthritis Versus the Use of Non-surgical Treatment: Randomized Clinical Trial and Comparison of Therapies for Medial Knee Osteoarthritis
Brief Title: MOTION Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moximed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP0011
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: 2:1 randomized controlled trial (RCT)
Who Masked: Outcomes Assessor
Masking Description: Randomization is programmed within the Electronic Data Capture system to ensure that the groups are unbiased and that the results are reliable, independent from the participant, investigator, and sponsor. The outcomes assessor remains independent from the participant, investigator and the sponsor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MISHA Knee System (Experimental): The MISHA Knee System is an extra-capsular knee implant intended to reduce loads on the medial knee. The implant consists of an absorber located between bases fixed with locking screws to the medial cortices of the distal femur and proximal tibia. The implant shares the load with the medial knee joint and articulating ball-and-sockets allow the device to accommodate the natural motions of the knee.
  Interventions: Device: MISHA Knee System
- Non-Surgical Treatment (Active Comparator): The non-surgical arm includes assist devices, physical conditioning, prescription or nonprescription medications, creams, vitamins, or supplements, intra-articular Injections, physical therapy and weight loss.
  Interventions: Other: Non-Surgical Treatment

INTERVENTIONS:
Device: MISHA Knee System — The MISHA Knee System is an extra-capsular knee implant intended to reduce loads on the medial knee. The implant consists of an absorber located between bases fixed with locking screws to the medial cortices of the distal femur and proximal tibia. The implant shares the load with the medial knee joint and articulating ball-and-sockets allow the device to accommodate the natural motions of the knee.
  Arms: MISHA Knee System
Other: Non-Surgical Treatment — The non-surgical arm includes assist devices, physical conditioning, prescription or nonprescription medications, creams, vitamins, or supplements, intra-articular Injections, physical therapy and weight loss.
  Arms: Non-Surgical Treatment

SUMMARY:
Prospective, multicenter, two-arm, 2:1 randomized controlled trial (RCT) comparing the benefits in subjects with medial knee osteoarthritis who are treated with either the MISHA Knee System or with non-surgical treatment.

This is the first randomized head-to-head study comparing outcomes from subjects treated with the MISHA Knee System.

ELIGIBILITY:
Key Inclusion Criteria:

1. Activity exacerbated knee pain isolated to the medial compartment and not global in nature
2. WOMAC pain ≥ 40
3. Failed to find relief in non-surgical treatment modalities

Key Exclusion Criteria:

1. Large medial osteophyte(s) or considerable extruded meniscus that may interfere with the placement or function of the device
2. Poor bone quality (e.g., bony erosion, osteopenia, osteoporosis)
3. Ligamentous instability
4. Active or recent knee infection
5. Inflammatory joint disease, including sequelae of viral infections
6. Suspected or documented allergy or hypersensitivity to cobalt, chromium, nickel or other metals
7. History of keloid, hypertrophic or contracture scaring
8. Propensity for restrictive scar formation or adhesions with prior procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
WOMAC Pain at 6 Months | 6 Months
  Improvement in WOMAC Pain in the MISHA arm compared to the non-surgical arm measured on the initial cohort who complete the 6-month follow-up visit

SECONDARY OUTCOMES:
WOMAC Function at 6 Months | 6 Months
  Improvement in WOMAC Function in the MISHA arm to the non-surgical arm measured on the fully enrolled population who complete the 6-month follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Rose S Weinstein, Study Director — Moximed
Locations (8):
- United States (8):
  - UC Davis Department of Orthopaedic Surgery, Davis, California
  - Scripps Clinic Jefferson, Oceanside, California
  - Rush University Medical Center, Chicago, Illinois
  - Genesis Orthopedics & Sports Medicine, Oak Brook, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone Health, New York, New York
  - Ohio State Jameson Crane Sports Medicine Institute, Columbus, Ohio
  - UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No